CLINICAL TRIAL: NCT01612416
Title: Comparison of Ganglion Cell and Retinal Nerve Fiber Layer Thickness in Primary Open Angle Glaucoma and Normal Tension Glaucoma With Spectral Domain OCT
Brief Title: Spectral Domain Optical Coherence Tomography Analysis for Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Penpe Gul Firat, Principal Investigator, Inonu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: TOTM 021
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: GLAUCOMA 1, OPEN ANGLE, D (Disorder)
Keywords: Ganglion Cell complex, Retinal Nerve Fiber Layer,Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal subjects (Sham Comparator)
  Interventions: Device: RS-3000 OCT measurements
- Primary open angle glaucoma (Active Comparator)
  Interventions: Device: RS-3000 OCT measurements
- Normal tension glaucoma (Active Comparator)
  Interventions: Device: RS-3000 OCT measurements

INTERVENTIONS:
Device: RS-3000 OCT measurements — Ganglion cell, retinal nerve fiber layer and retinal thickness measurements of normal subjects, primary open angle glaucoma and normal tension glaucoma patients using RS-3000 OCT RetinaScan
  Other Names: GCC and RNFL in Open Angle and Normal Tension Glaucoma.

SUMMARY:
The aim of this study is to examine whether there is a difference in macular ganglion cell complex thickness and retinal nerve fiber layer thickness in early-stage Primary open angle glaucoma and normal tension glaucoma with spectral domain OCT.

DETAILED DESCRIPTION:
Glaucoma is a progressive optic neuropathy characterized by gradual degeneration of neuronal tissue in which retinal ganglion cells (RGCs) are injured, leading to the loss of the visual field.Recent studies have separately demonstrated a reduction in the macular retinal thickness and in the retinal nerve fibers in both POAG and NTG.It has been demonstrated that in early stage NTG macular GCC thickness showed a strong correlation with thickness of the RNFL. However there have yet to be any reports regarding the comparison of macular thickness, ganglion cell complex and retinal nerve fiber layer between POAG and NTG with RS-3000 RetinaScan at early stage.

ELIGIBILITY:
Inclusion Criteria:

The POAG group inclusion criteria were;

* IOP higher than 21 mmHg before treatment on three different visits,
* Best corrected VA of 20/25 or better with a spherical equivalent within ±5 D and a cylinder correction within +3 D;
* An open angle confirmed by gonioscopy.
* Glaucomatous optic disc damage defined as by the presence of glaucomatous optic neuropathy like rim thinning (diffuse or local), cupping, notching, and a cup/disc ratio >0.2 with asymmetry.

NTG group were included if;

• They had the same optic disc and visual field criteria as for the POAG patients with the exception that their IOP was as ≤21 mmHg on three separate visits without any glaucomatous treatment.

The control group

* Who had no ocular disease
* Who had not undergone ocular surgery or laser procedures.
* With a normal anterior segment, open angles, and normal posterior segment findings also normal optic nerve head appearance in their ophthalmic examination.
* The IOP measurements were lower than 21 mmHg, and full-threshold 30-2 HFA were also within normal limits in the control group.

Exclusion Criteria:

* Subjects with any retinal disease, diabetes mellitus, or neurological disease or who had undergone ocular surgery and laser procedures.
* Subjects with pseudoexfoliation glaucoma and pigmentary glaucoma were excluded.

Ages: 28 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Ganglion cell complex, retinal nerve fiber layer and retinal thickness measurements of glaucoma patients using spectral domain OCT. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Penpe G Firat, M.D., Study Director — Assistant Professor; Selim Doganay, M.D, Principal Investigator — Professor; Ersan E Demirel, M.D., Principal Investigator — Resident; Cemil Colka, M.D., Study Chair — Associate Professor
Locations (1):
- Inonu University School of Medicine, Malatya, Turkey (Türkiye)

REFERENCES:
- [Background] Ojima T, Tanabe T, Hangai M, Yu S, Morishita S, Yoshimura N. Measurement of retinal nerve fiber layer thickness and macular volume for glaucoma detection using optical coherence tomography. Jpn J Ophthalmol. 2007 May-Jun;51(3):197-203. doi: 10.1007/s10384-006-0433-y. Epub 2007 Jun 7. PMID 17554482